CLINICAL TRIAL: NCT04434404
Title: Cardioprotection of Silymarin for Patients Received Anthracycline Chemotherapy
Brief Title: Evaluation of the Cardioprotective Effect of L-carnitine and Silymarin in Patients Receiving Anthracycline Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, hosny ahmed elewa, head of pharmacy practice department, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 32551/09/2018
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: anthracycline-containg chemotherapy; cardiotoxicity; breast cancer patients; slymarin; l-carnitine
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Carnitine; Tablets; Silymarin

STUDY DESIGN:
Intervention Model Description: This study was a parallel randomized (simple randomization; odd number took silymarin and even number took l carnitine) controlled prospective open label one.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): 33, patients in the control group received anthracycline-containing chemotherapy in a dose of 50 mg/m2 without cardioprotective agents
  Interventions: Drug: L-Carnitine 500Mg Oral Tablet
- L-carnitine group (Active Comparator): 25 patients received anthracycline-containing chemotherapy in a dose of 50 mg/m2 plus L-carnitine
  Interventions: Drug: L-Carnitine 500Mg Oral Tablet
- Silymarin group (Active Comparator): 25 patients received anthracycline-containing chemotherapy in a dose of 50 mg/m2 plus Silymarin140 mg
  Interventions: Drug: L-Carnitine 500Mg Oral Tablet

INTERVENTIONS:
Drug: L-Carnitine 500Mg Oral Tablet — eighty-three eligible patients were recruited 33, 25, and 25 patients in the control group, L-carnitine group, and, Silymarin group respectively, completed the study
  without cardioprotective agents in a dose of 50 mg/m2. L-carnitine group received anthracycline-containing chemotherapy in a dose of 50 mg/m2 plus L-carnitine 3 gm L-carnitine® capsules obtained from (MEPACO) was taken PO one day before chemotherapeutic cycle and 1gm /day during the following 21 days. Silymarin group received anthracycline-containing chemotherapy in a dose of 50 mg/m2 plus Silymarin as cardioprotective agent.140 mg (Legalon ® 140 mg capsule obtained from (MEDA). Silymarin was taken PO once daily after meals during the chemotherapeutic cycle. The treatment period was 6 months.
  Other Names: Silymarin

SUMMARY:
the study aim to protect patients received anthracyclines containing chemotherapy from cardiotoxcity induced by anthracyclines derivatives. by using L-carnitine and Silymarin for protection the heart from anthracyclines toxicities, and in addition its a comparitive study between L-carnitine and Silymarin.

DETAILED DESCRIPTION:
Aim: Anthracycline induced cardiotoxicity is the most common constrains of its use in treatment of various types of cancer. This study aimed to investigate benefits from adding L-carnitine and Silymarin compared to anthracycline chemotherapy alone in patients with cancer.

Methods: 83 patients were recruited from Clinical Oncology Department, Tanta University, Egypt, then prospectively randomized to receive their anthracycline containing therapeutic regimen, control group (n=33) or anthracycline plus L-carnitine, L-carnitine group (n=25), or anthracycline plus Silymarin, Silymarin group (n= 25). Blood samples were collected at begging and after 6 months to measure LDH, CK-MB, cTn I, Anticardiolipin IgG, Fe, ferritin and TIBC and % of saturation. % EF was documented. Data were statistically analyzed by ANOVA and paired t test. P <0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients receiving anthracycline chemotherapy in their protocol alone (without any cardioprotective agent),
* aged 20-60 and
* female patients were included.

Exclusion Criteria:

* patients with a history of heart failure, arrhythmia, history of cardiac catheterizations or, history of angina, uncontrolled hypertension and uncontrolled diabetes,
* patients with impaired liver function tests,
* previous anthracycline-containing regimens and any cardiotoxic chemotherapy regimens,
* previous history of chest wall irradiation.
* Brain metastasis,
* pregnant patients and
* patients who refused informed consent,

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — as all our participants were breast cancer patients
Enrollment: 83 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
The use of l-carnitine may be of use in extending the continuous use of anthracycline-containing chemotherapy | from the baseline untill 3 months
  addition of l-carnitine to the traditional therapy of breast cancer patients protocol containing anthracycline chemotherapy

SECONDARY OUTCOMES:
The use of silymarin may be of use in extending the continuous use of anthracycline-containing chemotherapy | from the baseline untill 3 months
  addition of silymarin to the traditional therapy of breast cancer patients protocol containing anthracycline chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Horus University, Damietta, Tanta City, Egypt

IPD SHARING:
Plan to Share IPD: No